CLINICAL TRIAL: NCT02290847
Title: Clinical Effectiveness Trial of In-Home Cognitive Processing Therapy for Combat-Related PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Duke University (Other); VA Boston Healthcare System (U.S. Federal Agency); South Texas Veterans Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC20140055H
Record Dates: First submitted 2014-11-05; First posted 2014-11-14 (Estimated); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Posttraumatic Stress Disorder; PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- In-Home Therapy (Active Comparator): Cognitive Processing Therapy (CPT-C) will be delivered to participants face to face in their homes by a certified therapist.
  Interventions: Behavioral: Cognitive Processing Therapy (cognitive only version; CPT-C)
- In-Office Therapy (Active Comparator): Cognitive Processing Therapy (CPT-C) will be delivered to participants face to face in a mental health clinic office setting by a certified therapist.
  Interventions: Behavioral: Cognitive Processing Therapy (cognitive only version; CPT-C)
- Telebehavioral Health (Active Comparator): Cognitive Processing Therapy (CPT-C) will be delivered to participants over the internet using video conferencing software by a certified therapist.
  Interventions: Behavioral: Cognitive Processing Therapy (cognitive only version; CPT-C)

INTERVENTIONS:
Behavioral: Cognitive Processing Therapy (cognitive only version; CPT-C) — CPT is a cognitive behavioral treatment for PTSD consisting of 12 one-hour sessions (Resick, Monson, & Chard, 2008; Resick & Schnicke, 1993). CPT is delivered in three phases: education, processing, and challenging. The manualized treatment focuses on challenging beliefs and assumptions related to the trauma, oneself, and the world.

SUMMARY:
The primary objective of this study is to evaluate the effectiveness of Cognitive Processing Therapy (cognitive only version; CPT-C) delivered using two different formats in the home setting for the treatment of combat-related PTSD as compared to conventional face-to-face CPT-C delivered in a mental health clinic. The study will include two different formats of in-home therapy: face-to-face in-home CPT-C and tele-behavioral health in-home CPT-C.

DETAILED DESCRIPTION:
The study will use a 3-arm equipoise-stratified randomization design (Lavori et al., 2001; Shalev et al., 2011) to evaluate the clinical effectiveness of CPT-C delivered in three formats: Face-to-Face In-Office (F2F-O), Face-to-Face In -Home (F2F-H), and Telebehavioral Health In -Home (TBH-H). The equipoise stratified design was specifically developed for clinical effectiveness trials involving multiple treatments that may not be appropriate for all research participants. The design will allow for complete randomization of those participants who are interested and eligible for all three treatment arms. It will also allow participants to opt out of one treatment arm if they are not interested or eligible for one of the arms. Without this provision a large proportion of the potential participants would be excluded from the study, seriously compromising external validity. Participants who elect to opt out of one arm will be randomized to one of the two remaining treatment arms. For example, the F2F-O treatment could be eliminated by those who are severely injured, home-bound, or seriously concerned about stigma, and they then would be randomized to receive one of the home-based CPT-C formats. The F2F-H treatment could be eliminated for participants who are uncomfortable with the idea of a mental health provider coming into their home. The telehealth arm could be opted out by veterans who are unable to use a computer, or cannot situate it in a private area.

The equipoise design will be used because a significant confound exists with the use of a completely randomized three-arm research design when all participants cannot be randomized to all arms. With a completely randomized design, participants must be willing to be randomized to all treatment arms or else they must be excluded. All participants willing to be randomized to all arms will occupy a universal donor stratum. The universal donor participants are randomized as in a completely randomized design, and they are able to participate in all statistical analyses. Participants that elect to opt out of one arm will enter a stratum comprising the remaining two arms, and they will be assigned at random to one of the two remaining arms. These participants may participate (along with those in the universal donor stratum) only in statistical analyses that compare arms to which they could have been randomized. By making a choice, each participant assigns himself or herself to a stratum, which consists of all the options that he or she finds equally acceptable. In this design, those who are unable to attend clinic will be randomized to one of the in-home arms. Those who are able to attend clinic will be given the option to reject any one of the three treatments. The randomization plan defines four strata (i.e., those who accept randomization to all three arms and those who reject one of the three treatments). Analyses will be done pairwise using only participants who accepted randomization to two or three treatments, and it will include stratum and the stratum-by-treatment interaction as design effects. Note that this design is the only way to include an in-clinic arm and a sample of participants who are unwilling or unable to be randomized to in-clinic treatment.

Specific Aims. The overall aim of the project is to conduct a 3-group randomized clinical trial to evaluate the clinical effectiveness of CPT-C delivered in three formats: (1) Face-to-Face In-Home CPT-C; (2) Face-to-Face In-Office CPT-C; and (3) Tele-Behavioral Health In-Home CPT-C.

Objective 1: Conduct a randomized clinical trial to evaluate the effectiveness of CPT-C delivered in three formats: (1) Face-to-Face In-Home CPT-C (F2F-H); (2) Face-to-Face In-Office CPT-C (F2F-O); and (3) Tele-Behavioral Health In-Home CPT-C (TBH-H) employing equipoise-stratified randomization.

Hypothesis 1: CPT-C delivered in F2F-H format will be more effective for the treatment of PTSD (symptom reduction below diagnostic threshold on the CAPS-5) than F2F-O & TBH-H.

Hypothesis 2: CPT-C delivered in F2F-H format will result in greater improvement in secondary outcomes (depression, alcohol consumption, marital and family functioning) than F2F-O & TBH-H.

Objective 2: Determine if standard F2F-O CPT-C can be enhanced and delivered to special populations (seriously injured, home-based rehab, rural living, severe avoidance) with in-home therapies.

Hypothesis 3: In-home therapies (F2F-H and TBH-H) will result in lower perceived stigma of seeking mental health care and higher treatment adherence (session attendance; out-of-session assignment completion; dose of therapy) compared to mental health clinic-based therapy.

Hypothesis 4: Participants who opt to participate in the in-home therapies (i.e., decline F2F-O) will have higher levels of treatment satisfaction than those in the F2F-O treatment arm.

ELIGIBILITY:
Inclusion Criteria

* Adult male and female active duty military and Veterans, with any previous military deployment seeking treatment for PTSD
* Person has experienced a Criterion A event that is a specific combat-related event or high magnitude operational experience that occurred during a military deployment. The diagnosis of PTSD may be indexed to that event or to another Criterion A event.
* Diagnosis of PTSD determined by the Clinician-Administered PTSD Scale - Interview - Version 5 (CAPS-5).
* Speak and read English.
* Participants taking psychotropic medications agree to work with their prescriber to remain on stable doses of any prescribed psychotropic medications for the duration of the intervention and through the first follow-up assessment as much as possible and as medically indicated.
* Patient must reside within a 45-mile radius of the UTHSCSA STRONG STAR offices in San Antonio.
* To participate in telemedicine study arm, participants must have access to a computer with a high definition display, high speed internet access, and USB port for installation of the HD telemedicine camera, OR be willing to use STRONG STAR equipment with necessary specifications for the duration of the telemedicine treatment phase.

  * The computer must be located in a private location where the participant will be able to control access during treatment encounters (ensuring their privacy and confidentiality).
  * The computer must be accessible enough to the participant to allow for the frequency and required number of encounters for the CPT intervention.
  * The computer must have high speed internet access (e.g., cable modem, USB, T1/T2 connection).
  * If a firewall is present on the participant's computer system, the participant needs to be able to arrange for access control to the system to allow the telepresence encounter to occur (i.e., they must either be able to open ports through the firewall or know someone who can arrange this for them).
  * The computer must be equipped with speakers or a standard headphone jack to allow access to audio output from the encounter (i.e., to be able to hear the therapist talking to them).
  * Telemedicine will be mediated by the Cisco C20 Quickset Telepresence System, an encrypted and could-based system. Because encounters are cloud-based, any participant can use the system if they have a computer and web-browser capable of processing most modern commercial internet services. Computer operating system will not matter.

Exclusion Criteria

* Current suicide or homicide risk meriting crisis intervention that is a higher priority than study participation.
* Endorsement of items pertaining to violence, arrest, probation, domestic abuse, or other issues that might suggest study staff would be at risk entering the home to deliver therapy as identified as part of the demographics.
* Alcohol and/or substance use that would prevent the participant from engaging in therapy.
* Active psychosis.
* Moderate to severe brain damage (as determined by the inability to comprehend the baseline screening questionnaires), as such individuals may be unable to fully benefit from the cognitive intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2014-09-19 (Actual); Primary Completion 2019-05-14 (Actual); Study Completion 2019-11-06 (Actual)

PRIMARY OUTCOMES:
PTSD Check List - DSM-5 (PCL-5), to assess change in PTSD symptomatology from baseline throughout treatment and at multiple follow up points | Baseline, Weekly during therapy (6 time points), 1 month Post-tx follow up, 2 Month Follow-Up, 3 Month Follow-Up, 4 Month Follow-Up, 5 Month Follow-Up, 6 Month Follow-Up
  The PCL-5 is a 20-item self-report measure based upon the DSM-5 criteria for PTSD that evaluates how much participants have been bothered by PTSD symptoms in the past month as a result of a specific life event. Each item of the PCL-5 is scored on a five point scale ranging from 0 "not at all") to 4 ("extremely).
Clinician-Administered PTSD Scale - 5 (CAPS-5); to assess change in PTSD symptomatology and/or diagnosis from baseline to multiple follow up points | Baseline, 1-month Post-tx Follow-Up, 3-month Follow-Up, 6-month Follow-Up
  The CAPS-5 is a structured interview that assesses the DSM-5 criteria for PTSD (Weathers et al., 2013). Each item is rated on a severity scale ranging from 0 (Absent) to 4 (Extreme) and combines information about frequency and intensity for each symptom. Validation studies are nearly complete to establish the psychometric properties of the CAPS-5. This interview is very similar to its predecessor, the CAPS for DSM-IV, which has been considered the gold standard for evaluating PTSD (Weathers, Keane, & Davidson, 2001). In addition to reflecting diagnostic changes for PTSD in DSM-5, the CAPS-5 differs from the CAPS in that frequency and intensity ratings for each symptom are no longer scored separately, so the severity rating for each item determines whether a symptom is present or not. Subscale scores are calculated by summing severity scores for items in the following PTSD symptom clusters: re-experiencing, avoidance, negative alterations in cognitions and mood, and hyperarousal.

CONTACTS AND LOCATIONS:
Overall Officials: Alan Peterson, PhD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- Strong Star, San Antonio, Texas, United States

REFERENCES:
- [Derived] Moring JC, Dismuke-Greer CE, Resick PA, Young-McCaughan S, Ortman J, McGeary C, Straud CL, Mackintosh MA, Acierno R, Rauch SAM, Morland LA, Peterson AL. Cost-effectiveness of evidence-based psychotherapies for PTSD: An examination of different treatment delivery modalities. Psychol Serv. 2026 Jan 26. doi: 10.1037/ser0001010. Online ahead of print. PMID 41587192
- [Derived] Moring JC, Peterson AL, Straud CL, Ortman J, Mintz J, Young-McCaughan S, McGeary CA, McGeary DD, Litz BT, Macdonald A, Roache JD, Resick PA, For The Strong Star Consortium. The interactions between patient preferences, expectancies, and stigma contribute to posttraumatic stress disorder treatment outcomes. J Trauma Stress. 2023 Dec;36(6):1126-1137. doi: 10.1002/jts.22982. Epub 2023 Oct 26. PMID 37883128
- [Derived] McGeary CA, Morland LA, Resick PA, Straud CL, Moring JC, Sohn MJ, Mackintosh MA, Young-McCaughan S, Acierno R, Rauch SAM, Mintz J, McGeary DD, Wells SY, Grubbs K, Nabity PS, McMahon CJ, Litz BT, Velligan DI, Macdonald A, Mata-Galan E, Holliday SL, Dillon KH, Roache JD, Peterson AL. Impact and efficiency of treatment across two PTSD clinical trials comparing in-person and telehealth service delivery formats. Psychol Serv. 2024 Feb;21(1):73-81. doi: 10.1037/ser0000774. Epub 2023 Jun 22. PMID 37347913
- [Derived] Peterson AL, Mintz J, Moring JC, Straud CL, Young-McCaughan S, McGeary CA, McGeary DD, Litz BT, Velligan DI, Macdonald A, Mata-Galan E, Holliday SL, Dillon KH, Roache JD, Bira LM, Nabity PS, Medellin EM, Hale WJ, Resick PA. In-office, in-home, and telehealth cognitive processing therapy for posttraumatic stress disorder in veterans: a randomized clinical trial. BMC Psychiatry. 2022 Jan 17;22(1):41. doi: 10.1186/s12888-022-03699-4. PMID 35038985